CLINICAL TRIAL: NCT01081756
Title: An Open, Randomized, Comparative Study Using Recombinant Human Chorionic Gonadotrophin (rhCG, Ovidrel®) in the Induction of Final Follicle Maturation and Early Luteinization in Chinese Women Undergoing in Vitro Fertilization and Embryo Transfer (IVF/ET)
Brief Title: A Study Using Recombinant Human Chorionic Gonadotrophin (rhCG, Ovidrel®) in the Induction of Final Follicle Maturation and Early Luteinization in Chinese Women Undergoing in Vitro Fertilization and Embryo Transfer (IVF/ET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Medical Director, Serono Singapore, an affiliate of Merck KGaA, Darmstadt, Germany.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP-25346
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2010-03

CONDITIONS: Infertility
Keywords: Reproductive technology; Assisted; recombinant human chorionic hormone (r-hCG)
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Chorionic Gonadotropin; Ovidrel; Profasi

ARMS (2):
- Subjects treated with r-hCG (Experimental): Subjects treated with r-hCG
  Interventions: Drug: r-hCG
- Subjects treated with urinary hCG (Active Comparator): Subjects treated with urinary hCG
  Interventions: Drug: Urinary-hCG

INTERVENTIONS:
Drug: r-hCG — r-hCG (250 mcg) injection subcutaneously (s.c.) or intramuscularly (i.m.)
  Other Names: Ovitrelle or Ovidrel
  Arms: Subjects treated with r-hCG
Drug: Urinary-hCG — Urinary hCG (10,000 IU) injection s.c. or i.m.
  Other Names: Profasi
  Arms: Subjects treated with urinary hCG

SUMMARY:
This was an open, randomized, comparative study using rhCG (Ovidrel) in the induction of final follicle maturation and early luteinization in Chinese female subjects undergoing IVF or ET.

DETAILED DESCRIPTION:
This was an open, randomized, comparative multicentric, phase III study to evaluate the safety and efficacy of rhCG in comparison with urinary hCG in the induction of final follicle maturation and early luteinization in 200 Chinese female subjects undergoing superovulation. The study was organized on an outpatient basis in subjects undergoing assisted reproductive technologies (ART). All subjects underwent pituitary down- regulation per each center's normal practice prior to and during stimulation of multiple follicular development. The subjects were randomized into 2 groups. One group received rhCG 250mcg and the other group received urinary hCG (Profasi®) 10,000IU. Each subject in both groups received a single injection of hCG when the follicular development was judged to be adequate. Oocytes were retrieved 36-38 hours after the hCG injection and fertilized in vitro. Not more than 3 embryos or 2 blastocysts were to be replaced. Progesterone was administered daily according to center's normal practice, starting after the oocyte pick up and continuing until a negative pregnancy test or for the first 3 weeks of pregnancy if the subject was pregnant. The subject was followed up and the treatment outcome (negative pregnancy test or pregnancy) was recorded.

A phase I sub-study to evaluate the pharmacokinetics of single subcutaneous (s.c.) administrations of rhCG was conducted on 24 healthy Chinese female subjects in China. The subjects were randomized into 3 groups. Each group received a single dose of 250mcg or 500mcg or 750 mcg of rhCG. Blood samples were collected at predetermined intervals after the injection. Human chorionic gonadotropin serum levels were measured with the Serono MAIAclone and the in vitro bioassay MA-10. Safety was assessed by the incidence and severity of adverse events (AEs), including multiple pregnancy and ovarian hyperstimulation syndrome (OHSS) and significant changes in laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Infertility regular ovulatory menstrual cycles;
* Early luteal phase serum levels:
* FSH≤ 10IU/l
* LH≤ 10IU/l
* PRL≤ 30ng/ml
* T≤ 50pg/ml
* Haematology, blood chemistry, urinalysis normal
* Both ovaries present
* < 3 previous ART cycles, no ART cycles for 2 menstrual cycles

Exclusion Criteria:

* With a poor response to gonadotrophin stimulation, such as ≤3 oocytes collected in any previous IVF cycle
* Any medical condition may interfere with the absorption, distribution, metabolism or excretion of the drug.
* Had previous severe ovarian hyperstimulation syndrome(OHSS)
* A body mass index (BMI) >25 kg/m2
* Any contraindication to being pregnant and/or carrying a pregnancy to term
* Extra-uterine pregnancy within the last 3 months
* A clinically significant systemic disease
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus
* Abnormal gynaecological bleeding of undetermined origin
* Known allergy or hypersensitivity to human gonadotrophin preparations
* Simultaneous participation in another clinical trial

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2003-12; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Number of oocyte retrieved | 36 hrs after hCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Huafei Li, Study Director — Serono Singapore
Locations (1):
- Peking University 3rd Hopistal, Beijing, China